CLINICAL TRIAL: NCT06700031
Title: Time on Feet After Hip Fracture Event - the TOFFEE Study
Brief Title: Time on Feet After Hip Fracture Event
Acronym: TOFFEE
Status: Not yet recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-07759-01
Record Dates: First submitted 2024-10-29; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Hip Fractures (ICD-10 72.01-72.2)
Keywords: hip fracture; mobilization; rehabilitation
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Inertial measurement unit — A sensor, an inertial measurement unit (IMU), will be attached to the thigh when the individual is on the postoperative ward and will be worn throughout the hospital stay. The IMU measures 7.9 x 3.2 x 0.8 cm and records body positions, movements, and gait parameters.

SUMMARY:
With simple technology investigators can map how long it takes for a patient with a hip fracture to be helped and encouraged to stand and walk in the days following the injury. A small sensor on the thigh can measure advanced data regarding movement patterns. The limited research results available show that patients spend too much time lying down or sitting, which can lead to poorer recovery, complications, and an increased risk of death. The project maps the current situation in orthopedic emergency care as well as in orthopedic geriatric care, which is provided in a modern building with single rooms and private bathrooms. In addition to better understanding the significance of different care models, the project aims to present baseline data that future intervention studies can use as control material. The project will also connect the activity level of the patients during the hospital stay with ongoing rehabilitation studies in community follow-up care.

DETAILED DESCRIPTION:
Purpose and Specific Objectives Can better diagnosis and prevention of inactivity after hip fractures improve outcomes for individuals and society? The goal is to measure how much individuals with hip fractures move during their hospital stay, to investigate the link between activity levels and complications such as thromboembolism, infections, and mortality, and to use inertial measurement units (IMU) to provide feedback to patients and healthcare providers.

Outcomes after frailty-related fractures remain poor, despite improved orthopedic surgical treatment. Every year, at least 50,000 people over the age of 65 in Sweden sustain a major fracture. Despite enhanced treatment and care, a fracture in older individuals often leads to permanent reductions in function and quality of life. Hip fractures are also associated with an increased risk of death. In addition to personal consequences, the many fractures have significant effects on healthcare and social elder care. Relatives are also affected. Falls are estimated to cost society over 14 billion kronor annually.

To improve recovery and avoid complications after a fracture, coworkers must think broadly and innovatively in healthcare. Given the rapid changes in lifestyle and socioeconomics, it is questionable whether healthcare providers can apply research findings based on previous generations to today's older adults, for example concerning physical activity.

A hip fracture is surgically treated so that the skeleton can withstand immediate weightbearing. However, patients spend too much time immobilized, according to the limited research available. This inactivity can lead to limited recovery, complications such as infections and thromboembolism, longer hospital stays, and an increased risk of death.

ELIGIBILITY:
Inclusion Criteria:

* Having an acute hip fractures and being admitted to either two wards with orthopedic standard care or to one with orthogeriatric care at Skane University Hospital, Malmö

Exclusion Criteria:

* Lack of standing ability prior to the fracture, defined as requiring a sling lift for transfer
* Skin disease that prevent the sensor from being attached (dry, flaky, or sore skin, or sensitivity to adhesive)
* Additional fractures besides the hip fracture or other injuries that reduce mobility (e.g., head or thoracic injuries)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with acute hip fractures regardless of age or cognitive status. The fracture should need surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-22 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Minutes in upright position per day | During hospital stay, an average of one week
  Sitting, standing or walking as measured by the IMU

SECONDARY OUTCOMES:
Complications within 30 days | 30 days from surgery
  Mortality and Incidence of infection or venous thromboembolism within 30 days
Association with type of fracture | During hospital stay, an average of one week
  Association between total time in upright position with type of fracture (intra- or extracapsular)
Association with type of surgical method | During hospital stay, an average of one week
  Association between total time in upright position with type of surgical method (hemiarthroplasty, total hip arthroplasty, internal fixation)
Association with duration of surgery | During hospital stay, an average of one week
  Association between total time in upright position with duration of surgery (min)
Association with age | During hospital stay, an average of one week
  Association between total time in upright position with age (years)
Association with sex | During hospital stay, an average of one week
  Association between total time in upright position with sex (male/female)
Association with comorbidities (ASA grade) | During hospital stay, an average of one week
  Association between total time in upright position with comorbidities measured by ASA grade (American society of anesthesiologists classification system)
Association with frailty (CFS) | During hospital stay, an average of one week
  Association between total time in upright position with frailty (CFS - Clinical Frailty Score)
Association with presence of dementia | During hospital stay, an average of one week
  Association between total time in upright position with presence of dementia (medical record information on ICD-code for dementia disease)

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Rogmark, PhD, Professor, Principal Investigator — Lund University; Eva Ekvall Hansson, PhD, Professor, Study Chair — Department of Health Sciences, Lund University
Locations (1):
- Dept. of Orthopaedics, Skane University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Swedish legislation is rigid on this point and request needs to be handled individually

REFERENCES:
- [Result] Moller U O, Fange A M, J K, D S, F F, Hansson E E. Modern technology against falls - A description of the MoTFall project. Health Informatics J. 2021 Apr-Jun;27(2):14604582211011514. doi: 10.1177/14604582211011514. PMID 34006139
- [Result] Howell DF, Malmgren Fange A, Rogmark C, Ekvall Hansson E. Rehabilitation Outcomes Following Hip Fracture of Home-Based Exercise Interventions Using a Wearable Device-A Randomized Controlled Pilot and Feasibility Study. Int J Environ Res Public Health. 2023 Feb 10;20(4):3107. doi: 10.3390/ijerph20043107. PMID 36833801